CLINICAL TRIAL: NCT07266753
Title: Oral Beta-lactams Versus Non-beta-lactamS for Treatment of Lower Extremity Osteomyelitis
Brief Title: Comparison of Oral Antibiotics For Bone Infections of the Leg and Foot
Acronym: OSTEO
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Michael Garron Hospital (Other)
Collaborators: University Health Network, Toronto (Other); The Ottawa Hospital Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDRU-INT-2024-004
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Osteomyelitis of Lower Extremities; Osteomyelitis - Foot; Osteomyelitis of the Foot
Keywords: Osteomyelitis; Bone Infection; Lower Extremity; Oral beta-lactams versus non-beta-lactams
MeSH Terms: conditions — Osteomyelitis | interventions — Monobactams

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Beta-Lactam Antibiotic (Experimental)
  Interventions: Drug: Oral Beta-Lactam Antibiotic
- Oral Non-Beta-Lactam Antibiotic (Active Comparator)
  Interventions: Drug: Oral Non-Beta-Lactam Antibiotic

INTERVENTIONS:
Drug: Oral Beta-Lactam Antibiotic — Participants in this arm are randomized to receive an oral antibiotic from the beta-lactam class (e.g., penicillins or cephalosporins) for the treatment of lower extremity osteomyelitis.
  Arms: Oral Beta-Lactam Antibiotic
Drug: Oral Non-Beta-Lactam Antibiotic — Participants in this arm are randomized to receive an oral antibiotic from the non-beta-lactam class (e.g., fluoroquinolones, lincosamides, sulfonamides) for the treatment of lower extremity osteomyelitis.
  Arms: Oral Non-Beta-Lactam Antibiotic

SUMMARY:
The goal of this clinical trial is to compare different classes of oral antibiotics (beta-lactam and non-beta-lactam antibiotics) for the treatment of bone infections of the leg and foot. The hypothesis is that oral beta-lactam antibiotics work as well as oral non-beta-lactam antibiotics to treat these infections. The first step is to assess whether it is possible to perform the trial by determining whether participants can be recruited and followed successfully. If the trial is proven to be possible, it will be expanded to ensure an answer to whether the two antibiotic classes work as well for the treatment of bone infections of the leg and foot.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (> 18 years old)
2. OM of the lower extremity (below the knee) as determined by the treating healthcare provider (clinically and/or radiographically)
3. Expected duration of treatment at least 28 additional days of antibiotic therapy for the infection episode, from the time of enrolment
4. Treating health care team has already transitioned or is willing to transition to oral antibiotic therapy for the remainder of the treatment duration

Exclusion Criteria:

1. Prior enrolment in the OSTEO trial
2. Already received more than 14 days of uninterrupted antibiotic treatment for this episode of OM
3. No beta-lactam or non-beta-lactam option due to any of:

   1. Allergy
   2. Suspected or confirmed antimicrobial resistance
   3. Medical contraindications
   4. Non-modifiable drug-drug interaction risk
4. Need to receive combination antibiotic therapy with both beta-lactam and non-beta-lactam, with the exception of metronidazole and rifampin
5. Prior antibiotic treatment for the same infection in the past 6 months
6. Known pregnancy, planning to become pregnant during the study period, or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1418 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Outcomes | 24 Weeks
  Cure (defined by meeting the criteria of: alive, not currently receiving antibiotics, no antibiotic switch from the assigned regimen and no surgical amputation)

SECONDARY OUTCOMES:
Secondary Effectiveness Outcomes | 24 Weeks
  The number of participant deaths.
Secondary Effectiveness Outcomes | 24 weeks
  Proportion of participants with an antibiotic switch (oral or IV)
Secondary Effectiveness Outcome | 24 weeks
  Number and level of amputations
Secondary Effectiveness Outcome | 24 weeks
  Number of debridement operations
Secondary Effectiveness Outcome | 24 weeks
  Proportion of participants receiving chronic antibiotics for infection suppression
Secondary Effectiveness Outcome | 24 weeks
  Total duration of antibiotics (oral and IV) for the initial treatment episode
Secondary Effectiveness Outcome | 24 weeks
  Number and type of antibiotic-related adverse events
Secondary Effectiveness Outcome | 24 weeks
  Quality of life measurement at 24 weeks (determined by EQ-5D questionnaire) The EQ-5D is a standardized instrument for measuring health-related quality of life. Scores range from 0 (worst possible health state) to 1 (best possible health state), with higher scores indicating better
Secondary Effectiveness Outcome | 24 weeks
  Wound colonization with a pathogen of interest
Secondary Effectiveness Outcome | 52 weeks
  Any positive clinical bacterial culture

OTHER OUTCOMES:
Feasibility Outcome | 24 weeks
  The proportion of potentially eligible participants approached for the trial who provide consent and are randomized (recruitment rate)
Feasibility Outcome | 24 weeks
  The proportion of participants who receive an initial dose of an antibiotic from the class to which they were randomly allocated (adherence rate)
Feasibility Outcome | 24 weeks
  The proportion of participants from whom the primary effectiveness outcome is obtained (complete outcome ascertainment rate).

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Ottawa Hospital, Ottawa, Ontario
  - Michael Garron Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided
Awaiting Research Ethics Board approval of the study.